CLINICAL TRIAL: NCT04525794
Title: BIOTRONIK- First-in-Human Assessment of the Safety and Clinical Performance of a Sirolimus Derivative-Coated Balloon (BRight DCB) in the Treatment of Subjects With de Novo Lesions in the Superficial Femoral and Proximal Popliteal Artery (BRight First Study)
Brief Title: BRight DCB First-in-Human Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik CRC Inc. (Industry)
Collaborators: Biotronik AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C1904
Record Dates: First submitted 2020-08-13; First posted 2020-08-25 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BRight DCB (Experimental)
  Interventions: Device: BRight DCB

INTERVENTIONS:
Device: BRight DCB — The BRight Drug-Coated Percutaneous Transluminal Angioplasty (PTA) Balloon catheter (BRight DCB) is intended for dilatation of de novo lesions in native superficial femoral or popliteal arteries with a simultaneous release of drug to the vessel wall as a secondary action to reduce occurrence of a restenosis of the treated vessel segment.

SUMMARY:
The primary aim of this clinical study is to assess the safety and clinical performance of the BRight drug-coated balloon (DCB) in the treatment of lower limb arteries stenosis in subjects with Peripheral Artery Disease (PAD).

The primary endpoint will be Late Lumen Loss (LLL) of the target lesion at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has provided written informed consent
2. The subject is willing to participate in the clinical investigation and to comply with the study procedures and follow-up visits
3. Lifestyle-limiting claudication or rest pain requiring treatment of superficial femoral (SFA) and/or proximal popliteal artery (PPA)
4. Rutherford-Becker Clinical Category of 2, 3 or 4
5. Target vessel reference diameter ≥5 mm and ≤ 6 mm (by visual estimation)
6. De novo lesion with >50% stenosis by operator visual estimate within the SFA and/or proximal popliteal arteries in a single limb.
7. Lesion must be located ≥ 1 cm below the Common Femoral Artery (CFA) bifurcation and terminate distally at ≥ 3 cm proximal to the knee joint (radiographic joint space)
8. Single lesion length ≤100 mm for de novo stenotic lesions, or ≤ 70 mm for occluded lesions (one long lesion or multiple serial lesions) by operator visual estimate. Note: Only 1 lesion per patient can be treated. Multiple serial lesions are allowed provided that they can be treated as a single lesion with one balloon.
9. Successful guidewire crossing of lesion.
10. After pre-dilatation, the target lesion is ≤ 30% residual stenosis with no flow limiting dissection and treatable with a single balloon
11. Inflow artery is patent, free from significant lesion stenosis (>50% stenosis considered significant) as confirmed by angiography.
12. Target limb with at least 1 patent (less than 50% stenosis) tibio-peroneal run-off vessel in the target limb confirmed at baseline. (Note: treatment of outflow disease is not permitted.)

Exclusion Criteria:

1. Females who are pregnant, lactating, or intended to become pregnant, or males intending to father children during the study
2. Subject under current medication known to affect CYP3A4 metabolism
3. Contraindication to dual anti-platelet therapy
4. Subject is receiving chronic anticoagulation therapy (e.g. low molecular weight heparin, warfarin, or novel direct oral anticoagulants (N(D)OACs)).
5. Known intolerance to study medications, Limus- like drug or contrast agents that in the opinion of the investigator could not be adequately pretreated
6. Current participation in an investigational drug or another device study
7. History of hemorrhagic stroke within 3 months
8. Patients with a history of Myocardial Infarction (MI) or thrombolysis within 30 days prior-index procedure
9. Previous or planned surgical or interventional procedure within 14 days before or 30 days after index procedure (successful treatment of the ipsilateral and contralateral iliac arteries is permitted prior to enrollment- contralateral iliac artery treatment with no drug eluting technology is allowed during the index procedure)
10. Prior endovascular treatment of the target lesion (e.g., POBA, DCB, BMS, DES, cutting balloons, scoring balloons, cryoplasty, thrombectomy, atherectomy, brachytherapy or laser devices)
11. Previous placement of a bypass graft proximal to the target lesion
12. Chronic renal insufficiency (eGFR < 30 mL/min within 72 hours prior to index procedure)
13. No normal proximal arterial segment in which duplex ultrasound velocity ratios could be measured.
14. Subject is unable to walk without assistance (e.g. walker, cane).
15. Subject is receiving immunosuppressant therapy.
16. Subject has known or suspected active infection at the time of the index procedure.
17. Subject has platelet count < 100,000/mm3 or > 700,000/mm3.
18. Subject has white blood cell (WBC) count < 3,000/mm3.
19. Subject is unable to tolerate blood transfusions because of religious beliefs or other reasons.
20. Subject has history of gastrointestinal hemorrhage requiring a transfusion within 3 months prior to the index procedure.
21. Life expectancy less than 12 months due to other comorbidities, that in the investigators opinion, could limit subject ability to comply with the study required follow-up visits/procedure and threaten the study scientific integrity
22. Treatment of the contralateral limb during the same procedure or within 30 days following the study procedure (exclusive of the iliac arteries, which can be treated prior to enrollment or during the index procedure if no drug eluting technology is used)
23. Non femoral vascular access
24. Target lesion would require treatment with more than one balloon
25. Known inadequate distal outflow
26. Acute or sub-acute thrombus in the target vessel
27. Aneurysmal target vessel
28. Use of adjunctive therapies (i.e. laser, atherectomy, cryoplasty, scoring/cutting balloon, brachytherapy) during the study procedure in the target lesion or target vessel
29. Presence of concentric calcification that precludes PTA pre-dilatation
30. Significant contralateral or ipsilateral common femoral disease that requires intervention during the index procedure
31. Persistent hemodynamically-significant stenosis following predilatation or residual stenosis of >30%, stent placement, or flow-limiting (Grade D or greater) dissection following pre-dilatation
32. In-stent restenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
Late Lumen Loss | 6 months post index procedure
  Late Lumen Loss, as measure by quantitative vascular angiography (QVA)

SECONDARY OUTCOMES:
Device success | during procedure
  Successful delivery, balloon inflation/deflation and retrieval of the intact trial device
Acute technical success | during procedure
  Successful vascular access and completion of the endovascular procedure and immediate achievement of a final residual diameter stenosis of ≤30% of the treated lesion by core laboratory assessed QVA on the completion angiography with no bailout stenting
Acute procedural success | 72 hours post index procedure
  Technical success without the occurrence of death, major target limb amputation, thrombosis of the target lesion, or clinically-driven TLR within 72 hours of the index procedure
Major Adverse Event (MAE) rate | 1, 6 and 12 months post index procedure
  MAE is a composite of device or procedure related death within 30 days post index procedure, major index limb amputation, cd TLR
Clinically-driven Target Lesion Revascularization (cd TLR) rate | 1, 6 and 12 months post index procedure
  cd TLR is defined as any repeat intervention of the target lesions or surgical bypass of the target vessel performed for restenosis > 50% or other complication involving the target lesion, after documentation of recurrent clinical symptoms of the patient.
Clinically-driven Target Vessel Revascularization (cd TVR) rate | 1, 6 and 12 months post index procedure
  cd TVR, defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel, after documentation of recurrent clinical symptoms of the patient.
All-cause of death rate | 1, 6 and 12 months post index procedure
Amputation (minor and major) rate | 1, 6 and 12 months post index procedure
  rate of amputation (minor and major)
Change in Rutherford Classification as compared to baseline | 1, 6 and 12 months post index procedure
  change in the Rutherford classification between baseline and follow-up
Change in resting target limb Ankle Brachial Index (ABI) as compared to baseline | 1, 6 and 12 months post index procedure
  change in ABI between baseline and follow-up
Target lesion Binary Restenosis | 1, 6 and 12 months post index procedure
  Defined as duplex ultrasound peak systolic velocity ratio (PSVR) > 2.5 (if DUS is completed) or angiographic assessment which suggests stenosis > 50% by QVA
Target lesion primary patency | 1, 6 and 12 months post index procedure
  Target lesion primary patency defined as duplex ultrasound peak systolic velocity ratio (PSVR) ≤ 2.5 (if DUS is completed) or angiographic assessment which suggests stenosis ≤ 50% by QVA and the absence of Clinically-driven TLR (adjudicated by a CEC)
Change in the Walking Impairment questionnaire (WIQ) as compared to baseline | 1, 6 and 12 months post index procedure
  change in WIQ between baseline and follow-up
Embolic event of the index limb | during procedure
  occurrence of embolic event as visualized on angiography

CONTACTS AND LOCATIONS:
Locations (7):
- Australia (4):
  - Prince of Wales Hospital, Randwick, New South Wales
  - Fiona Stanley Hospital, Perth
  - Royal Perth Hospital, Perth
  - Royal North Shore Hospital, Sydney
- Medical University Graz, Graz, Styria, Austria
- Klinikum Hochsauerland, Arnsberg, Germany
- Auckland City Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No